CLINICAL TRIAL: NCT01474590
Title: Efficacy and Safety Comparison of Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel Associated With 200 mg Doxycycline Capsules Versus Vehicle Gel Associated With Isotretinoin Capsules in the Treatment of Severe Acne
Brief Title: Efficacy & Safety Comparison of Epiduo With Doxycycline Versus Vehicle With Isotretinoin in the Treatment of Severe Acne
Acronym: POWER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD.03.SPR.29099
Record Dates: First submitted 2011-11-16; First posted 2011-11-18 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2017-08

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene, Benzoyl Peroxide Drug Combination; Doxycycline; Isotretinoin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epiduo/Tactuo + doxycycline 200mg (Experimental)
  Interventions: Drug: Epiduo/Tactuo; Drug: doxycycline 200mg
- Isotretinoin + vehicle gel (Active Comparator)
  Interventions: Other: vehicle gel; Drug: Isotretinoin

INTERVENTIONS:
Drug: Epiduo/Tactuo — topical to the face, once daily in the evening
  Arms: Epiduo/Tactuo + doxycycline 200mg
Other: vehicle gel — topical to the face, once daily in the evening
  Arms: Isotretinoin + vehicle gel
Drug: doxycycline 200mg — oral, 2 capsules once daily in the morning with aglass of water and with food
  Arms: Epiduo/Tactuo + doxycycline 200mg
Drug: Isotretinoin — oral, 0.5mg/kg/day for a period of four weeks, adjusted to 1 mg/kg/day for the four following months.
  Arms: Isotretinoin + vehicle gel

SUMMARY:
Non-inferiority, randomized, controlled, multi-center, investigator-blind, parallel-group comparison study in subjects with severe acne vulgaris on the face.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject of any race, aged 12 to 35 years inclusive
2. Subject weighing between 50 and 110 kg
3. Subject with severe acne (IGA at least 4), which in the opinion of the investigator is appropriate for treatment with oral isotretinoin (severe nodular acne, severe inflammatory acne, recalcitrant acne; all unresponsive to conventional first line therapies)
4. Subject with at least 5 nodules on the face

Exclusion Criteria:

1. Subject with clinically abnormal results to blood testings performed at screening
2. Subject with acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc.), pyoderma faciale, sinus tracks
3. Female subject who is pregnant, nursing or planning a pregnancy during the study
4. Subject with known history of hepatic and/or renal insufficiency, to be confirmed by blood testings
5. Subject with known metabolic or structural bone disease (for 12-17 years old population)
6. Subject with bowel disease and/or with hypervitaminosis A
7. Subject who presents with treated or untreated depression or has a history of depression including a family history of major depression
8. Subject with a wash-out period from baseline for topical treatment on the face less than : Corticosteroids, antibiotics, antibacterials, antiseptics, retinoids, other anti-inflammatory drugs or other acne treatments (2 weeks); Cosmetic procedures (1 week); Photodynamic therapy and laser therapy for acne (3 months)
9. Subject with a wash-out period from baseline for systemic treatment less than: Corticosteroids, antibiotics (4 weeks),Progesterone for contraception (3 months); Spironolactone(3 months); Other acne treatments (6 months);Cyproterone acetate(6 months)

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 266 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Tan, Principal Investigator — Windsor Clinical Research Inc.
Locations (25):
- Canada (25):
  - Galderma investigational site, Ajax
  - Galderma investigational site, Barrie
  - Galderma investigational site, Calgary
  - Galderma investigational site, Edmonton
  - Galderma investigational site, Greater Sudbury
  - Galderma investigational site, Halifax
  - Galderma investigational site, Hamilton
  - Galderma investigational site, Markham
  - Galderma investigational site, Montreal
  - Galderma investigational site, Newmarket
  - Galderma investigational site, Oakville
  - Galderma investigational site, Oshawa
  - Galderma investigational site, Peterborough
  - Galderma investigational site, Québec
  - Galderma investigational site, Richmond Hill
  - Galderma investigational site, Saint-Hyacinthe
  - Galderma investigational site, Saskatoon
  - Galderma investigational site, St. John's
  - Galderma investigational site, Surrey
  - Galderma investigational site, Toronto
  - Galderma investigational site, Vancouver
  - Galderma investigational site, Waterloo
  - Galderma investigational site, Windsor
  - Galderma investigational site, Winnipeg
  - Galderma investigational site, Woodbridge

REFERENCES:
- [Derived] Tan J, Humphrey S, Vender R, Barankin B, Gooderham M, Kerrouche N, Audibert F, Lynde C; POWER study group. A treatment for severe nodular acne: a randomized investigator-blinded, controlled, noninferiority trial comparing fixed-dose adapalene/benzoyl peroxide plus doxycycline vs. oral isotretinoin. Br J Dermatol. 2014 Dec;171(6):1508-16. doi: 10.1111/bjd.13191. Epub 2014 Oct 28. PMID 24934963

RESULTS

PARTICIPANT FLOW:
Groups:
- Epiduo/Tactuo + Doxycycline 200mg: Epiduo/Tactuo + doxycycline 200mg: Epiduo gel: topical to the face, once daily in the evening Doxycycline: oral, 2 capsules a day. The capsules should be taken with a glass of water and with food either as a single dose or in two divided doses during the day.
- Isotretinoin + Vehicle Gel: Isotretinoin + vehicle gel: Vehicle gel: topical to the face, once daily in the evening Isotretinoin: oral, 0.5mg/kg/day for a period of four weeks, adjusted to 1 mg/kg/day for the four following months.
Period: Overall Study
Arm/Group | Epiduo/Tactuo + Doxycycline 200mg | Isotretinoin + Vehicle Gel
Started | 133 | 133
Completed | 105 | 116
Not Completed | 28 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epiduo/Tactuo + Doxycycline 200mg | Isotretinoin + Vehicle Gel | Total
Number analyzed (Participants) | 133 | 133 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.5 (5.0) | 19.3 (4.5) | 19.4 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 115 | 112 | 227
Region of Enrollment [Number; unit: count of participants]
  Canada | 133 | 133 | 266
IGA [Number; unit: count of participants] — the global severity assessment is outlined as per below:
  Investigator's Global Assessment (IGA)
  score
  0. Clear: Residual hyperpigmentation and erythema may be present
  1. Almost Clear A few scattered comedones and a few small papules
  2. Mild Some comedones and some papules and pustules. No nodules present
  3. Moderate Many comedones, papules and pustules. One nodule may be present
  4. Severe Covered with comedones, numerous papules and pustules and few nodules may be present
  5. Very severe Highly inflammatory acne covering the face; with nodules present
  count of participants
    4 | 118 | 115 | 233
    5 | 15 | 18 | 33
nodule counts [Mean (Standard Deviation); unit: nodules] | 8.0 (3.6) | 7.6 (2.5) | 7.8 (3.1)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome is Overall Success, a Composite Endpoint Including Efficacy and Safety Measurements
Description: Overall success is reached when the 2 following criteria are fulfilled :
  1. Overall efficacy: reduction of at least 75% of number of nodules at the end of treatment
  2. Safe treatment: Absence of any listed safety issues
Time Frame: 20 weeks
Measure: Number; unit: count of participants
Arm/Group | Epiduo/Tactuo + Doxycycline 200mg | Isotretinoin + Vehicle Gel
Number analyzed (Participants) | 133 | 133
count of participants | 85 | 73

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Epiduo/Tactuo + Doxycycline 200mg | Isotretinoin + Vehicle Gel
Serious Adverse Events (participants affected / at risk) | 0/133 | 1/133
Other Adverse Events (participants affected / at risk) | 25/133 | 66/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epiduo/Tactuo + Doxycycline 200mg (N=133) | Isotretinoin + Vehicle Gel (N=133)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epiduo/Tactuo + Doxycycline 200mg (N=133) | Isotretinoin + Vehicle Gel (N=133)
dry skin (Skin and subcutaneous tissue disorders) | 25 (31) | 43 (56)
skin irritation (Skin and subcutaneous tissue disorders) | 14 (17) | 7 (8)
headache (Nervous system disorders) | 12 (14) | 11 (12)
lip dry (Gastrointestinal disorders) | 9 (9) | 66 (72)
nausea (Gastrointestinal disorders) | 14 (14) | 5 (5)
vomiting (Gastrointestinal disorders) | 12 (14) | 2 (2)
naospharyngitis (Infections and infestations) | 15 (17) | 14 (17)
UPTRI (Upper Tract Respiratory Infection) (Infections and infestations) | 9 (10) | 13 (16)
cheilitis (Gastrointestinal disorders) | 2 (2) | 32 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other